CLINICAL TRIAL: NCT04787328
Title: A Single-arm, Open-Label, Multicenter Phase II Study to Evaluate the Efficacy and Safety of HA121-28 Tablets in Patients With Medullary Thyroid Carcinoma (MTC)
Brief Title: A Study of HA121-28 Tablets in Patients With Medullary Thyroid Carcinoma (MTC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA122-CSP-003
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Medullary Thyroid Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA121-28 tablets (Experimental): Patients will receive HA121-28 tablets at 450 mg once daily (QD) for 21 days on a 28-day treatment cycle.
  Interventions: Drug: HA121-28 tablets

INTERVENTIONS:
Drug: HA121-28 tablets — HA121-28 450 mg, po, QD×21 days, every 4 weeks (28 days)

SUMMARY:
This is a single-arm, open-label, multicenter study designed to evaluate the preliminary antineoplastic activity, safety and tolerability of HA121-28 tablets administered orally in patients with medullary thyroid cancer (MTC).

DETAILED DESCRIPTION:
A total of approximately 30 patients with MTC will be enrolled. The patients will undergo a 3 weeks-on and 1week-off treatment scheme with HA121-28 tablets 450 mg orally once daily in the 28-day cycle until disease progression or intolerable toxic reaction, whichever occurs first. During the administration of HA121-28 tablets, vital signs, physical examination, ECOG performance status, hematology and chemistry test, ECG, adverse events and concomitant drugs will be evaluated every four weeks, an additional ECG will be observed two weeks after the first dose, calcitonin and pregnancy test will be performed every 8 weeks. CT for tumor assessment will be performed every 8 weeks for the first year, and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to participate in the clinical trial and sign the informed consent;
2. Men and women aged ≥18 years;
3. Histologically confirmed unresectable locally advanced or metastatic MTC with at least one measurable lesion per RECIST1.1;
4. Evidence of disease progression within 12 months prior to signing informed consent;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1;
6. Laboratory test results must meet the following criteria: Absolute neutrophil count (ANC) ≥1.5 x 10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin (Hb) ≥90 g/L; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) (in patients with liver metastasis ≤5.0 x ULN); Total bilirubin ≤ 1.5 x ULN; Serum creatinine≤ 1.5 x ULN；Prothrombin time (PT) and activated Partial Thromboplastin Time (APTT) ≤ 1.5 x ULN；
7. Left ventricular ejection fraction (LVEF)≥50% in echocardiogram；
8. Male and female subjects of childbearing potential must agree to take effective contraception during the treatment period and for 6 months after the last dose of study medication;
9. Female participants must have negative results of serum/urine pregnancy test within 7 days prior to enrollment and must not be breastfeeding.

Exclusion Criteria:

1. Previous treatment with selective RET inhibitor, such as blu-667, loxo-292, etc.;
2. Patients who had participated in other clinical trials and received the treatment within 4 weeks prior to enrollment;
3. Systemic anti-tumor treatment such as small molecule targeted drugs, cytotoxic drugs, immunotherapy and radiotherapy within 4 weeks of the first dose of the study drug, or local palliative radiotherapy for pain relief within 2 weeks;;
4. Patients who cannot swallow or have chronic diarrhea (except for those induced by MTC) and intestinal obstruction, or other factors which may affect the administration and absorption of the study drug;
5. History of other malignancies within the past 5 years or currently suffering from other malignancies, except for cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumor;
6. Patients who meet one of the following criteria: 1) Corrected QT (QTc) ≥450 ms (corrected using Fridericia's formula (QTcF): QTcF = QT/(RR^0.33)); 2) Any clinically significant abnormalities of rhythm, conduction or morphology in the resting electrocardiogram (ECG) requiring therapeutic intervention;
7. Urine protein≥2+ and urine protein > 1.0 g/24h;
8. Known severe concomitant and/or uncontrolled diseases, including but not limited to: 1)Uncontrolled hypertension (systolic pressure ≥150 mmHg or diastolic pressure ≥100 mmHg, after treatment); 2)Significant cardiovascular and cerebrovascular events, arterial or venous fistulae thrombotic events, myocardial infarction, congestive heart failure (NYHA classification ≥2) or severe ventricular arrhythmia within 6 months of the first dose of the study drug; 3) Liver cirrhosis, decompensated liver disease; 4) Renal failure required hemodialysis or peritoneal dialysis; 5) History of human immunodeficiency, including HIV positive, or other acquired/congenital immune deficiency diseases, or history of organ or bone marrow transplantation; 6) Uncontrolled pericardial effusion, pleural effusion or ascites;7） interstitial pneumonia required steroid therapy or severe infection required systemic treatment, which is judged not suitable for the study by the investigator;
9. Patients with spinal cord, meningeal and brain metastases (except for stable symptomatic or asymptomatic brain metastases);
10. Ongoing adverse events>grade 1 due to any previous treatment at the time of enrollment (except for hair loss and pigmentation);
11. Patients who have undergone major surgery or have not recovered from invasive operation within 4 weeks prior to initiation of study treatment;
12. Patients with bleeding diathesis (such as active peptic ulcer) or treated with anticoagulants or vitamin K antagonists, such as warfarin, heparin or their analogues;
13. Known active Hepatitis B or Hepatitis C virus infection: HBsAg positive with HBV DNA higher than the lower limit of detection range of the site, or HCV antibody positive with HCV RNA higher than the lower limit of detection range of the site);
14. Patients with known history of neurological or psychiatric disorders, including epilepsy or dementia;
15. Not suitable for the study assessed by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first, assessed up to 60 months
  assessed approximately every 8 weeks or 12 weeks based on the treatment cycle

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression, assessed up to 60 months
  assessed approximately every 8 weeks or 12 weeks based on the treatment cycle
Duration of response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first, assessed up to 60 months
  assessed approximately every 8 weeks or 12 weeks based on the treatment cycle
Overall survival (OS) | From date of randomization until date of death from any cause, assessed up to 60 months
  assessed approximately every 12 weeks
Disease control rate (DCR) | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first, assessed up to 60 months
  assessed approximately every 8 weeks or 12 weeks based on the treatment cycle
Changes in blood calcitonin | From date of randomization until the date of first documented progression or date of death from any cause, or date of death from any cause,whichever came first, assessed up to 60 months
  assessed approximately every 8 weeks
Adverse events incidence | From date of randomization until the date of death from any cause, assessed up to 60 months
  assessed approximately every 4 weeks
Plasma drug concentration | From date of randomization until the date of first documented progression or date of death from any cause, wihichever came first, assessed up to 60 months
  assessed approximately every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Master, Study Director — CSPC ZhongQi Pharmaceutical Technology Co., Ltd.
Locations (13):
- China (13):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Province Tumor Hospital, Zhengzhou, Henan
  - Jiangsu province tumor hospital, Nanjing, Jiangsu
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No